CLINICAL TRIAL: NCT04039386
Title: Psychosocial Interventions for Young Adults With Hip Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michael C Willey (Other)
Responsible Party: Sponsor-Investigator, Michael C Willey, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1111
Record Dates: First submitted 2019-05-16; First posted 2019-07-31 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hip Dysplasia; Hip Pain Chronic; Hip Osteoarthritis; Hip Arthritis; Psychosocial Problem
Keywords: Hip Pain; Hip Instability; Hip Impingement; Cognitive Based Therapy; Psychosocial Conditions
MeSH Terms: conditions — Hip Dislocation; Osteoarthritis, Hip | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cell Phone Based Cognitive Based Therapy (Experimental): Young adults with hip pain
  Interventions: Device: Cell Phone Based Cognitive Based Therapy (Pacifica App)
- Placebo (Placebo Comparator): Young adults with hip pain
  Interventions: Other: Control

INTERVENTIONS:
Device: Cell Phone Based Cognitive Based Therapy (Pacifica App) — Cell phone application that provides support for individuals with psychosocial conditions.
  Arms: Cell Phone Based Cognitive Based Therapy
Other: Control — Subjects in the control group will receive standard care.
  Other Names: Standard Care
  Arms: Placebo

SUMMARY:
Psychosocial conditions are common in young adults with hip pain including depression, anxiety, pain catastrophizing, and narcotic use. The incidence of these conditions is not well defined. Interventions to optimize psychosocial conditions with non-surgical or surgical treatments has not been investigated. The goal of this project is to determine the incidence of psychosocial conditions in the young adult population with hip pain and determine if cognitive based therapy can improve clinical outcomes in these individuals.

DETAILED DESCRIPTION:
Over the last 3 decades there has been a drastic increase in the number of joint preservation surgeries performed for pre-arthritic hip conditions in the United States. Despite advances in surgical technique and the understanding of the biomechanics of impingement and dysplasia, failure rates range from 5-20% at early follow up, and can be even higher with continued monitoring. These failures are often attributed to the presence of pre-operative osteoarthritis, increased age, or unaddressed structural deformity. The influence of psychosocial factors on surgical and rehabilitative outcomes has been recognized in multiple populations, but has largely been ignored in individuals with hip pathology, in spite of growing recognition by clinicians as to how psychosocial factors may contribute to patient outcomes. Previous investigations have demonstrated poor mental health is associated with pre-operative narcotic use and lower physical function. Further, the investigators have identified certain psychiatric diagnoses as independent factors associated with failure of hip arthroscopy. Addressing these often complex psychosocial issues using cognitive based therapy has been successful in improving outcomes across a range of medical conditions. Further investigation into the incidence of these psychosocial conditions, their contributions to surgical and non-surgical outcomes, and interventions for mental health optimization need to be performed in musculoskeletal medicine, specifically in the developing field of hip preservation surgery. The goal of this project is to (1) understand the burden of maladaptive psychosocial traits in young adult patients with hip pain, and (2) reduce pain, decrease narcotic use, and improve physical function through psychosocial intervention delivered concomitantly during physical therapy. The investigators seek to maximize outcomes of individuals with non-arthritic hip dysfunction by addressing maladaptive behaviors so subjects can more effectively participate in rehabilitative treatment, and potentially, avoid the need for surgical management.

ELIGIBILITY:
Inclusion Criteria:

* We will enroll young adults (15-39) presenting to one of several physical therapy and orthopedic practices in the state of Iowa for treatment of nonarthritic hip pain.
* Chief complaint of hip pain or dysfunction, and a diagnosis of a nonarthritic hip condition including labral tear, femoroacetabular impingement (FAI), snapping hip, femoral anteversion or dysplasia.

Exclusion Criteria:

* Exclusion criteria will include age <15 or >40 years
* Difficulty with written English
* Treatment for alternative conditions such as trochanteric bursitis, hip dislocation, avascular necrosis or fracture.

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in level of Depression (DASS-21) | 8 weeks
  Assessed using the Depression Anxiety Stress Scale (DASS-21) electronically administered patient reported outcome questionnaire
  * General adult population average total score: 9.43 (standard deviation (SD) 9.66), out of a total possible score of 63 points,
  * Indication of significant difference from normative data: Average score >1 SD above the General adult population average total score
  * General adult population average depression sub scale score: 2.83 (SD 3.87)
  * Values above 9.03 points in the depression subsection score correlate with clinical depression and generalized anxiety disorders
  * A change of 3.86 or more points in the depression subscore reliably represents clinical improvement.
Changes in level of Depression (PROMIS) | 8 weeks
  Assessed using the Patient Reported Outcome Measures Information (PROMIS): Depression. An electronically administered patient reported outcome questionnaire
  * Normative T-score generated from US adult population data: mean 50 (SD 10).
  * For this study, an average T-score <40 would be considered significantly different compared to normative values.
  * The minimally important difference (MID) of 3.0-3.1 calculated from research in nonoperative treatment of knee osteoarthritis will be representative of clinical improvement at eight weeks.
Changes in level of Anxiety (DASS-21) | 8 weeks
  Assessed using the Depression Anxiety Stress Scale (DASS-21) electronically administered patient reported outcome questionnaire
  * General adult population average total score: 9.43 (SD 9.66)
  * An average total score >1 SD above the mean would be considered significantly different from normative data
  * General adult population average anxiety subscale scores: 1.88±2.95
  * Average anxiety subsection score above 6.27 correlate with clinical depression and generalized anxiety disorders
  * A change of 3.85 or more points in the anxiety subscore reliably represents clinical improvement.
Changes in level of Anxiety (PROMIS) | 8 weeks
  Assessed using the Patient Reported Outcome Measures Information (PROMIS): Anxiety. An electronically administered patient reported outcome questionnaire
  * Normative T-score generated from US adult population data: mean 50 (SD 10).
  * For this study, an average T-score <40 would be considered significantly different compared to normative values.
  * The minimally important difference (MID) of 2.3 to 3.4 calculated from research in nonoperative treatment of knee osteoarthritis will be representative of clinical improvement at eight weeks.
Changes in level of Stress (DAAS-21) | 8 Weeks
  Assessed using the Depression Anxiety Stress Scale (DASS-21) electronically administered patient reported outcome questionnaire
  * General adult population average total score: 9.43 (SD 9.66)
  * An average total score >1 SD above the mean would be considered significantly different from normative data
  * General adult population average stress subscale scores: 4.73±4.20
  * Average stress subsection score above 12.27 correlate with clinical depression and generalized anxiety disorders
  * A change of 4.90 or more points in the anxiety subscore reliably represents clinical improvement.
Evaluating the presence and severity of Kinesiophobia | 8 weeks
  Assessed via the Shortened Tampa Scale for Kinesiophobia (TSK-11) electronically administered patient reported outcome questionnaire
  * The survey is a 11-question test scored from 11-44, where higher scores indicate increasing fear of movement.
  * A value of 11 is presumed in a nonpainful population.
  * Adults with chronic musculoskeletal pain undergoing outpatient chronic pain therapy report an average TSK score of 30.4 (+/- 6.6).
  * Successful evaluation of Kinesiophobia will be indicated if increases in TSK-11 scores are found to be significantly associated with increased pain and decreased physical function (HOOS, PROMIS-PI, PROMIS-PB, PROMIS-PF) or increased self-reporting of opioid use.
  * The finding of no significant association, but increased presence of maladaptive features compared to normative data for US adolescents would also be considered a successful finding.
Evaluation of Resiliency | 8 weeks
  Assessed via The Brief Resiliency Scale (BRS) electronically administered patient reported outcome questionnaire
  * An 8 question survey scored from 1-5 points
  * The average score for US adults age 24-34 is 3.2 (SD 0.7)
  * A statistically significant lower Grit score would be >1SD below this average value.
  * Successful evaluation of Grit will be indicated if increases in GRIT-S scores are found to be significantly associated with increased pain and decreased physical function (HOOS, PROMIS-PI, PROMIS-PB, PROMIS-PF) or increased self-reporting of opioid use.
  * The finding of no significant association, but increased presence of maladaptive features compared to normative data for US adolescents would also be considered a successful finding.
Evaluation of Grit | 8 weeks
  Assessed via The Short Grit Scale (GRIT-S) electronically administered patient reported outcome questionnaire
  * A 6-question test with low resiliency defined as a score of <3.00.
  * Prior descriptive studies indicate an average score of 3.57 (SD 0.76) for young adults age 19.8±3.0 years.
  * Statistically significant lower resilience would be >1SD below this average value.
  * Successful evaluation of Resiliency will be indicated if increases in GRIT-S scores are found to be significantly associated with increased pain and decreased physical function (HOOS, PROMIS-PI, PROMIS-PB, PROMIS-PF) or increased self-reporting of opioid use.
  * The finding of no significant association, but increased presence of maladaptive features compared to normative data for US adolescents (for those tests where this data exists) would also be considered a successful finding.
Evaluating the presence and severity of Pain Catastrophizing | 8 weeks
  Assessed via Pain Catastrophizing Scale (PCS) electronically administered patient reported outcome questionnaire
  * Scored on a 13 point scale.
  * Normative average values from a population of adults adults age 42.2 (17-63 years) with low back pain: mean 20.90 (SD 12.5),
  * Successful evaluation of Pain Catastrophization will be indicated if increases in PCS scores are found to be significantly associated with increased pain and decreased physical function (HOOS, PROMIS-PI, PROMIS-PB, PROMIS-PF) or increased self-reporting of opioid use.
  * The finding of no significant association, but increased presence of maladaptive features compared to normative data for US adolescents would also be considered a successful finding.
Evaluating Self-Efficacy | 8 weeks
  Assessed via The General Self-Efficacy Scale (GSE) electronically administered patient reported outcome questionnaire
  * 10-question test, scored from 10-40, with lower scores representing low self efficacy.
  * Average US adult values: 29.48 (SD 5.13)
  * Successful evaluation of Self-Efficacy will be indicated if increases in GSE scores are found to be significantly associated with increased pain and decreased physical function (HOOS, PROMIS-PI, PROMIS-PB, PROMIS-PF) or increased self-reporting of opioid use.
  * The finding of no significant association, but increased presence of maladaptive features compared to normative data for US adolescents would also be considered a successful finding.
Evaluating the presence and severity of Alcohol Use Disorders | 8 weeks
  Assessed via Alcohol Use Disorders Identification Test (AUDIT) electronically administered patient reported outcome questionnaire
  * A 10-question test with a threshold score >7 considered "AUDIT-positive", indicating risky or hazardous alcohol use behavior.
  * National data suggests 15-20% of US 14-18 year olds screen positive
  * Successful evaluation of Alcohol Use Disorders will be indicated if increases in AUDIT scores are found to be significantly associated with increased pain and decreased physical function (HOOS, PROMIS-PI, PROMIS-PB, PROMIS-PF) or increased self-reporting of opioid use.
  * The finding of no significant association, but increased presence of maladaptive features compared to normative data for US adolescents would also be considered a successful finding.
Changes in Physical Function (PROMIS) | 8 weeks
  Measured via the following electronically administered patient reported outcome questionnaires.
  * PROMIS: Physical Function (PF)
  * Normative T-score generated from US adult population data: mean 50 (SD 10).
  * For this study, an average T-score <40 would be considered significantly different compared to normative values.
  * The minimally important difference (MID) of 1.9 - 2.2 calculated from research in nonoperative treatment of knee osteoarthritis will be representative of clinical improvement at eight weeks.
Changes in Physical Function (HOOS) | 8 weeks
  Measured via the following electronically administered patient reported outcome questionnaires.
  * The Hip disability and osteoarthritis outcome score (HOOS)
  * Scored from 0-100
  * Increasing score represent better function.
  * Average scopres for hip preservation patients prior to surgery is well established
Reduced Opioid Use | 8 weeks
  Measured via self reported opioid use after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Scott, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No